CLINICAL TRIAL: NCT01140815
Title: A Prospective, Single-Center, Randomized Study Comparing the Functional Performance of the Journey Deuce Bicompartmental With the Genesis II Total Knee System
Brief Title: Functional Performance of the Journey Deuce Bicompartmental Versus the Genesis II Total Knee System
Acronym: Deuce
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anderson Orthopaedic Research Institute (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Nancy Parks, Knee Project Director, Anderson Orthopaedic Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AORI2010-0103
Record Dates: First submitted 2010-05-28; First posted 2010-06-10 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Bicompartmental Knee Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Total (Active Comparator): The Smith and Nephew Total Knee System
  Interventions: Device: Total Knee Replacement
- Deuce (Experimental): The Journey Deuce Bicompartmental Knee System
  Interventions: Device: Deuce

INTERVENTIONS:
Device: Total Knee Replacement — Smith and Nephew Total Knee Replacement
  Arms: Total
Device: Deuce — Smith and Nephew Bicompartmental Knee Replacement
  Arms: Deuce

SUMMARY:
The objectives of this study are to assess the safety and effectiveness of the Journey Deuce Bicompartmental Knee System at 4-6 weeks, 4 months, 1 year, and 2 years when compared to total knee replacement using the Genesis II Total Knee System. The hypothesis is that the Journey Deuce Bicompartmental Knee System is as safe and effective as the Genesis II Total Knee System at the 2-year. The null hypothesis is that there is no difference between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient presents with non-inflammatory degenerative joint disease of the medial and patellofemoral compartments requiring a unilateral knee replacement.
* Patient is 30 to 65 years of age, inclusive.
* Patient is willing to consent to participate in the study by signing and dating an IRB-approved consent form.
* Patient plans to be available for follow-up through 2 years postoperative.

Exclusion Criteria:

* Patient is known to have insufficient femoral or tibial bone stock resulting from conditions such as cancer, distal femoral/proximal tibial osteotomy, significant osteoporosis or metabolic bone disorders.
* Patient is immunosuppressed, has an autoimmune disorder, or an immunosuppressive disorder (i.e. chronic condition characterized by markedly inhibited ability to respond to antigenic stimuli.) Examples of such conditions include patients who are on immunosuppressive therapy (corticosteroid hormones in large amounts, cytotoxic drugs, antilymphocytic serum or irradiation in large doses) or patients with acquired immunodeficiency syndrome (AIDS).
* Patient has inflammatory arthritis (e.g. rheumatoid arthritis)
* Patient has BMI > 35.
* Patient has had major knee surgery in the past i.e. HTO, unicondylar knee replacement, failed fracture fixation.
* Patient has an active infection, local or systemic.
* Patient has physical, emotional or neurological conditions that would compromise the patient's compliance with postoperative rehabilitation and follow-up (e.g.: drug or alcohol abuse, serious mental illness, or general neurological conditions such as Parkinson, Multiple sclerosis, etc.).
* Patient has ACL deficiency in the study knee.
* Patient has hip arthritis and/or replacement.
* Patient has lateral compartment disease.
* Patient is pregnant or plans to become pregnant during the course of the study.
* Patient is on workman's compensation.
* Patient has a known sensitivity to materials in the device.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard A. Engh, MD, Principal Investigator — AORI
Locations (1):
- Anderson Orthopaedic Research Institute, Alexandria, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited preoperatively in a clinical setting between 2007-2010.
Pre-assignment Details: Patients with only unicondylar arthritis were excluded and underwent unicondylar arthroplasty. Patients with arthritis in the lateral compartment were excluded and underwent total knee arthroplasty.
Period: Overall Study
Arm/Group | Total | Deuce
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Preoperative osteoarthritis of the knee in medial and patellofemoral joints. BMI less than or equal to 35, Age less than or equal to 65. No previous knee surgery.
Groups:
- Total (Control): The Smith and Nephew Total Knee System
  Total Knee Replacement: Smith and Nephew Total Knee Replacement
- Deuce (Study): The Journey Deuce Bicompartmental Knee System
  Deuce: Smith and Nephew Bicompartmental Knee Replacement
- Total: Total of all reporting groups
Arm/Group | Total (Control) | Deuce (Study) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Full Range); unit: years] | 58.3 [45 to 65] | 60.3 [53 to 65] | 59.3 [45 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 6 | 9 | 15
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Body Mass Index [Mean (Full Range); unit: lbs/square inches] | 30 [25 to 35] | 28.8 [23 to 34] | 29.2 [23 to 35]
Knee Score [Mean (Full Range); unit: units on a scale] | 50 [15 to 78] | 52.7 [20 to 90] | 51.3 [15 to 90]

OUTCOME MEASURES:

1. Primary Outcome: 2-Year Knee Society Score
Description: Knee Society Clinical Rating System (KSS) provides for separate knee pain and patient functional assessment scores. Scale of 0-100 with higher values representing a better score.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: units on a scale 0-100
Arm/Group | Total | Deuce
Number analyzed (Participants) | 25 | 25
units on a scale 0-100 | 91.3 (9.6) | 94.2 (5.6)

2. Primary Outcome: 6-Week Knee Society Score
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale 0-100
Arm/Group | Total | Deuce
Number analyzed (Participants) | 25 | 25
units on a scale 0-100 | 75 (15.7) | 83.3 (15)

3. Primary Outcome: 4-Month Knee Society Score
Description: as for outcome 1
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale 0-100
Arm/Group | Total | Deuce
Number analyzed (Participants) | 25 | 25
units on a scale 0-100 | 87.1 (10.2) | 91.3 (9)

4. Primary Outcome: 1-year Knee Society Score
Description: as for outcome 1
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale 0-100
Arm/Group | Total | Deuce
Number analyzed (Participants) | 25 | 25
units on a scale 0-100 | 88.6 (14.6) | 91.7 (9.2)

5. Secondary Outcome: 6-Week X-rays
Description: Knee Society Roentgenographic Evaluation and Scoring System will assess alignment; any evidence of loosening as indicated primarily by radiolucencies > 2mm; evidence of surface wear or particulate debris generation as indicated by early osteolysis, implant migration, or other clinical or radiographic abnormalities. Number of participants with these radiographic abnormalities by X-ray at 6 weeks are reported.
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Total | Deuce
Number analyzed (Participants) | 25 | 25
participants | 0 | 0

6. Secondary Outcome: 4-month X-rays
Description: Knee Society Roentgenographic Evaluation and Scoring System will assess alignment; any evidence of loosening as indicated primarily by radiolucencies > 2mm; evidence of surface wear or particulate debris generation as indicated by early osteolysis, implant migration, or other clinical or radiographic abnormalities. Number of participants with these radiographic abnormalities by X-ray at 4 months are reported.
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Total | Deuce
Number analyzed (Participants) | 25 | 25
participants | 0 | 0

7. Secondary Outcome: 1-year X-rays
Description: Knee Society Roentgenographic Evaluation and Scoring System will assess alignment; any evidence of loosening as indicated primarily by radiolucencies > 2mm; evidence of surface wear or particulate debris generation as indicated by early osteolysis, implant migration, or other clinical or radiographic abnormalities. Number of participants with these radiographic abnormalities by X-ray at 1 year are reported.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Total | Deuce
Number analyzed (Participants) | 25 | 25
participants | 2 | 3

8. Secondary Outcome: 2-year X-rays
Description: Knee Society Roentgenographic Evaluation and Scoring System will assess alignment; any evidence of loosening as indicated primarily by radiolucencies > 2mm; evidence of surface wear or particulate debris generation as indicated by early osteolysis, implant migration, or other clinical or radiographic abnormalities. Number of participants with these radiographic abnormalities by X-ray at 2 years are reported.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Total | Deuce
Number analyzed (Participants) | 25 | 25
participants | 6 | 4

9. Secondary Outcome: 2-year Patient Surveys
Description: Serial patient evaluation of function will be assessed using the Oxford Knee Outcome Questionnaire. The Oxford Questionnaire consists of 12 questions, each with a value of 0 (bad) to 4(good). The results are summed for a total score of 0(bad) to 48(good).
Time Frame: 2 years
Population: Patients who were not revised within 2 years and were able to complete a questionnaire did so.
Measure: Mean (Full Range); unit: units on a scale 0-48
Arm/Group | Total (Control) | Deuce (Study)
Number analyzed (Participants) | 23 | 23
units on a scale 0-48 | 41 [24 to 48] | 43 [32 to 47]

10. Secondary Outcome: 6-week Functional Testing
Description: A timed Functional Assessment Test, gait analysis, and balance testing for lower extremity motor function will be performed. Fewer seconds in the result indicates faster performance, which is a positive result.
Time Frame: 6 weeks
Population: Patients who were not revised and were able to make an appointment and complete the testing did so.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Total (Control) | Deuce (Study)
Number analyzed (Participants) | 24 | 25
seconds | 36.5 (10.7) | 35.1 (15.6)

11. Secondary Outcome: 4-month Functional Testing
Description: as for outcome 10
Time Frame: 4 months
Population: Patients who were not revised and were able to make an appointment and complete the testing did so.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Total (Control) | Deuce (Study)
Number analyzed (Participants) | 24 | 24
seconds | 25.5 (3.7) | 26.7 (4.8)

12. Secondary Outcome: 1-year Functional Testing
Description: as for outcome 10
Time Frame: 1 year
Population: Patients who were not revised and were able to make an appointment and complete the testing did so.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Total (Control) | Deuce (Study)
Number analyzed (Participants) | 23 | 22
seconds | 25 (5.6) | 23.9 (3.4)

13. Secondary Outcome: 2-year Functional Testing
Description: as for outcome 10
Time Frame: 2 years
Population: Patients who were not revised and were able to make an appointment and complete the testing did so.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Total (Control) | Deuce (Study)
Number analyzed (Participants) | 23 | 23
seconds | 25.1 (2.9) | 23.3 (3.7)

ADVERSE EVENTS:
Arm/Group | Total (Control) | Deuce (Study)
Serious Adverse Events (participants affected / at risk) | 1/25 | 3/25
Other Adverse Events (participants affected / at risk) | 3/25 | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (Control) (N=25) | Deuce (Study) (N=25)
Revision knee arthroplasty (Surgical and medical procedures) | 1 | 3 — Implant revised for loosening
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (Control) (N=25) | Deuce (Study) (N=25)
Knee stiff (Musculoskeletal and connective tissue disorders) | 3 | 1 — Manipulation of the knee under anesthesia for stiffness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days